CLINICAL TRIAL: NCT03627845
Title: A Phase 1, Single-Center, Randomized, Double-Blind, Placebo-Controlled Single-Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of PHP-303 in Healthy Subjects
Brief Title: A Study of Safety, Tolerability, and Pharmacokinetics of Single Doses of PHP-303 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: pH Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PHP-303-N101
Record Dates: First submitted 2018-07-31; First posted 2018-08-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2019-03

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): PHP-303, single oral dose, up to 6 ascending dose cohorts
  Interventions: Drug: PHP-303
- Placebo (Placebo Comparator): Placebo, single oral dose, up to 6 ascending dose cohorts
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PHP-303 — Investigational drug
  Arms: Experimental
Other: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled single ascending dose (SAD) study designed to evaluate the safety, tolerability, and pharmacokinetics (PK) of PHP-303 in healthy volunteer subjects. Within each ascending dose cohort, subjects will be randomized in a 3:1 ratio to receive PHP-303 or placebo. The primary objective is to establish the safety and tolerability of orally-administered PHP-303.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, ≥ 18 to ≤ 55 years of age.
* In good general health having no clinically significant diseases in medical history or evidence of clinically significant findings on physical examination, vital signs, laboratory results, and/or ECG at Screening, in the opinion of an Investigator.
* Willing to forego other forms of experimental treatment during the study.

Exclusion Criteria:

* Any clinically significant condition that, in the opinion of an Investigator, could preclude the safe participation of the subject in the study or would prevent the subject from meeting the study requirements.
* Major surgery in the 6 months preceding Screening.
* Clinically-significant abnormal laboratory parameters.
* Positive urine drug test for alcohol, cotinine, and/or drugs of abuse (cocaine, tetrahydrocannabinol, amphetamines, methamphetamines, or benzodiazepines) at Screening or on admission to the study site.
* Electrocardiographic Fridericia's corrected QT interval (QTcF) interval > 450 msec for males and > 470 msec for females, or any other clinically significant electrocardiographic abnormality.
* Blood pressure results > 150 mmHg systolic or > 95 mmHg diastolic
* Female subject who is pregnant (positive pregnancy test at the Screening Visit or on admission to the study site), lactating, or planning to become pregnant during the study period or within 3 months after the final dose of study medication.
* History of drug or alcohol abuse or dependence within 1 year prior to Screening.
* History of cigarette smoking within 3 months of Screening.
* Known intolerance to lactose.
* Regular use of prescription drugs within 14 days of the first administration of study drug or non-prescription (over-the-counter) drugs within 7 days of the first administration of study drug or unwilling to abstain from prohibited medications through the end of study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2020-01-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single oral dose of PHP-303 - Incidence of Adverse Events | Up to 9 weeks
  Assess the number of patients with adverse events
Safety and tolerability of single oral dose of PHP-303 - number of patients with abnormal ECG | Up to 9 weeks
  Number of patients with clinically significant change from baseline in standard 12 lead ECG parameters
Safety and tolerability of single oral dose of PHP-303 - blood pressure | Up to 9 weeks
  Number of patients with clinically significant change from baseline in systolic and diastolic blood pressure
Safety and tolerability of single oral dose of PHP-303 - heart rate | Up to 9 weeks
  Measured as number of heart beats per minute
Safety and tolerability of single oral dose of PHP-303 - body temperature | Up to 9 weeks
  Measurement of oral body temperature
Safety and tolerability of single oral dose of PHP-303 - respiratory rate | Up to 9 weeks
  Measured by number of breaths per minute
Plasma concentration of single oral dose of PHP-303 - AUC | Up to 9 weeks
  Area under the curve
Plasma concentration of single oral dose of PHP-303 - Cmax | Up to 9 weeks
  Maximum observed concentration
Plasma concentration of single oral dose of PHP-303 - t1/2 | Up to 9 weeks
  Determination of half-life

CONTACTS AND LOCATIONS:
Overall Officials: Brian Roberts, MD, Study Chair — pH Pharma Inc
Locations (1):
- Vince & Associates Clinical Research, Inc., Overland Park, Kansas, United States